CLINICAL TRIAL: NCT03700515
Title: Exosome Proteomics to Detect Eyrthropoietin (EPO) Use in Athletes
Brief Title: Exosome Proteomics to Detect EPO
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Morten Hostrup, PhD (Other)
Collaborators: University of Tasmania (Other)
Responsible Party: Sponsor-Investigator, Morten Hostrup, PhD, Associate Professor, University of Copenhagen
Organization: University of Copenhagen (Other)
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Basic Science
Other Study IDs: EPO-EXO
Record Dates: First submitted 2018-09-27; First posted 2018-10-09 (Actual); Last update posted 2019-09-25 (Actual); Status verified 2019-09

CONDITIONS: Healthy
Keywords: EPO
MeSH Terms: interventions — Erythropoietin

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (3):
- Placebo (Placebo Comparator): Saline infusion
  Interventions: Drug: Placebo
- EPO (Experimental): Erythropoetin infusion (9 IU/kg)
  Interventions: Drug: Erythropoietin
- EPO II (Experimental): Erythropoetin infusion (20 IU/kg)
  Interventions: Drug: Erythropoietin

INTERVENTIONS:
Drug: Erythropoietin — Subjects receive weekly infusions of EPO
  Arms: EPO; EPO II
Drug: Placebo — Subjects receive weekly infusions of saline
  Arms: Placebo

SUMMARY:
The role of exosomes in cell signalling has only recently been appreciated and is a hugely exciting and rapidly growing area, and combined with LC-MS/MS proteomics, can overcome traditional barriers to proteomics in doping applications. To our knowledge, no research has yet been undertaken to explore whether the highly promising combination of exosome proteomics has utility for rhEPO detection. The applications are extensive; the diagnostic value of differentially regulated proteins could be further validated against the existing IEF EPO WADA accredited tests using samples collected during this study, used to study altitude hypoxia versus exogenous EPO administration (WADA current targeted research 2017), investigated as a platform approach to ESA and HIF agents more generally, as well as facilitate development of direct ELISA high throughput tests.

ELIGIBILITY:
Inclusion Criteria:

* VO2max of at least 55+/-2 for men and 50+/-2 for women
* BMI between 18 and 27
* Resting hematocrit of less than 46%

Exclusion Criteria:

* Chronic disease deemed by the medical doctor to affect the outcome
* Competitive athlete subject to doping control
* Use of other prescription medicine deemed by the medical doctor to interact with the study drug
* Allergy or otherwise unacceptable side effects toward the study drug
* Smoker
* Pregnancy

Ages: 18 Years to 45 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 72 (Estimated)
Dates: Start 2019-09-04 (Actual); Primary Completion 2020-10-15 (Estimated); Study Completion 2020-10-15 (Estimated)

PRIMARY OUTCOMES:
Blood proteome enrichment pathway analysis in GO annotation | At baseline and after week 3 of treatment
  Change in enrichment (measured in blood and assessed using GO annotation)

SECONDARY OUTCOMES:
Blood markers of iron | At baseline and after week 3 of treatment
  Change in blood markers of iron homeostasis

CONTACTS AND LOCATIONS:
Locations (1):
- August Krogh Building, Copenhagen, Denmark

IPD SHARING:
Plan to Share IPD: Undecided